CLINICAL TRIAL: NCT06697132
Title: Modified Antegrade Stenting in Laparoscopic Pediatric Pyeloplasty; an Optimized Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelghany, lecturer, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N-443-2023
Record Dates: First submitted 2024-08-25; First posted 2024-11-20 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-08

CONDITIONS: UPJ - Ureteropelvic Obstruction
MeSH Terms: conditions — Multicystic renal dysplasia, bilateral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Modified antegrade stenting in laparoscopic pediatric pyeloplasty (Experimental)
  Interventions: Procedure: laparoscopic dismembered pyeloplasty

INTERVENTIONS:
Procedure: laparoscopic dismembered pyeloplasty — Modified antegrade stenting in laparoscopic pediatric pyeloplasty

SUMMARY:
Background and Rationale For decades, the use of transanastomotic stents following dismembered pyeloplasty has been controversial. However classically, many surgeons used to insert an indwelling DJ stent to secure the ureteropelvic anastomosis. During the laparoscopic pyeloplasty, the DJ can be inserted using different approaches. Neither of these approaches has absolute benefits , nor is free from drawbacks.

Objective: Whether the retrograde or antegrade approach of stenting is superior in laparoscopic pyeloplasty remains a great controversy. Each technique has its advantages and disadvantages. We tried in this study to optimize the way of stenting, taking the advantages of both approaches and avoiding their disadvantages.

DETAILED DESCRIPTION:
Objective: Whether the retrograde or antegrade approach of stenting is superior in laparoscopic pyeloplasty remains a great controversy. Each technique has its advantages and disadvantages. We tried in this study to optimize the way of stenting, taking the advantages of both approaches and avoiding their disadvantages.

Methods: Between March 2013 and August 2021, 75 patients less than 15 years of age candidate for laparoscopic pyeloplasty were included in the study. All cases were done by the same surgeon in our institute. At first, a retrograde study was done, and an open-tip ureteric catheter was inserted just below the pelviureteric junction. Putting the ureteric catheter just below the pelviureteric junction makes the whole procedure easier. After proper dissection, the anterior wall of the pelvis is incised and continuing the ureteric spatulation on its lateral aspect. Before the complete division of the ureter, the first stitch is taken between the angle of ureteric spatulation and the lower angle of the pelvis. After completing the posterior wall anastomosis, a guide wire is introduced through the ureteric catheter, grasped gently, and pulled out through the uppermost port, and the ureteric catheter is then removed. With the proximal end of the guide wire passing through the upper port and its distal end coming outside the urethra, the DJ is passed in an antegrade manner while pulling on the urethral catheter balloon to close the bladder neck.

ELIGIBILITY:
Inclusion Criteria:

* all pediatric patients (less than 15 years old) candidates for laparoscopic dimembered pyeloplasty.

Exclusion Criteria:

* • patiens who have any contraindications for pneumoperitoneum.

  * Children more than 15 y old
  * Children undergoing stentless pyeloplasty
  * Patients undergoing pyeloplasty other than dismembered type.

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
operative and post operative complication rate | one year

IPD SHARING:
Plan to Share IPD: No